CLINICAL TRIAL: NCT03375164
Title: Systemic Gene Delivery Phase I/IIa Clinical Trial for Duchenne Muscular Dystrophy Using rAAVrh74.MHCK7.Micro-dystrophin (microDys-IV-001)
Brief Title: A Gene Transfer Therapy Study to Evaluate the Safety of Delandistrogene Moxeparvovec (SRP-9001) in Participants With Duchenne Muscular Dystrophy (DMD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRP-9001-101; 2021-000077-83 (EudraCT Number)
Record Dates: First submitted 2017-12-04; First posted 2017-12-15 (Actual); Results first posted 2024-05-23 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne; Gene Therapy; DMD; Dystrophin; Pediatric; Gene-Delivery; Gene Transfer Therapy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: Delandistrogene Moxeparvovec (Experimental): Participants will receive a Single IV infusion of delandistrogene moxeparvovec on Day 1.
  Interventions: Genetic: delandistrogene moxeparvovec
- Cohort B: Delandistrogene Moxeparvovec (Experimental): Participants will receive a Single IV infusion of delandistrogene moxeparvovec on Day 1.
  Interventions: Genetic: delandistrogene moxeparvovec

INTERVENTIONS:
Genetic: delandistrogene moxeparvovec — Single IV infusion of delandistrogene moxeparvovec.
  Other Names: SRP-9001; delandistrogene moxeparvovec-rokl; ELEVIDYS

SUMMARY:
This study was an open-label single-dose gene transfer therapy study evaluating the safety of delandistrogene moxeparvovec intravenous (IV) administration in boys with DMD. This study was originally designed to consist of 12 patients across 2 Cohorts. Cohort A would have included participants ages 3 months to 3 years, and Cohort B included participants ages 4 to 7 years old. No participants were enrolled in Cohort A.

ELIGIBILITY:
Inclusion Criteria:

* Cohort A participants: 3 months to 3 years of age, inclusive
* Cohort B participants: 4 to 7 years of age, inclusive
* Definitive diagnosis of DMD based on documented clinical findings and prior genetic testing.
* Ability to cooperate with motor assessment testing.
* Cohort A participants: No previous treatment with corticosteroids.
* Cohort B participants: Stable dose equivalent of oral corticosteroids for at least 12 weeks prior to screening and the dose is expected to remain constant (except for potential modifications to accommodate changes in weight) throughout the first year of the study.
* Cohorts A & B: A frameshift mutation contained between exons 18 and 58 (inclusive).

Exclusion Criteria:

* Exposure to gene therapy, investigational medication, or any treatment designed to increase dystrophin expression within protocol specified time limits.
* Abnormality in protocol-specified diagnostic evaluations or laboratory tests.
* Presence of any other clinically significant illness, medical condition, or requirement for chronic drug treatment that in the opinion of the Investigator creates unnecessary risk for gene transfer.

Other inclusion or exclusion criteria could apply.

Ages: 3 Months to 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Zaidman CM, Proud CM, McDonald CM, Lehman KJ, Goedeker NL, Mason S, Murphy AP, Guridi M, Wang S, Reid C, Darton E, Wandel C, Lewis S, Malhotra J, Griffin DA, Potter RA, Rodino-Klapac LR, Mendell JR. Delandistrogene Moxeparvovec Gene Therapy in Ambulatory Patients (Aged >/=4 to <8 Years) with Duchenne Muscular Dystrophy: 1-Year Interim Results from Study SRP-9001-103 (ENDEAVOR). Ann Neurol. 2023 Nov;94(5):955-968. doi: 10.1002/ana.26755. Epub 2023 Sep 7. PMID 37539981
- [Derived] Mendell JR, Sahenk Z, Lehman K, Nease C, Lowes LP, Miller NF, Iammarino MA, Alfano LN, Nicholl A, Al-Zaidy S, Lewis S, Church K, Shell R, Cripe LH, Potter RA, Griffin DA, Pozsgai E, Dugar A, Hogan M, Rodino-Klapac LR. Assessment of Systemic Delivery of rAAVrh74.MHCK7.micro-dystrophin in Children With Duchenne Muscular Dystrophy: A Nonrandomized Controlled Trial. JAMA Neurol. 2020 Sep 1;77(9):1122-1131. doi: 10.1001/jamaneurol.2020.1484. PMID 32539076
- See also: SRP-9001-101 Plain Language Study Summary — https://www.sarepta.com/sites/sarepta-corporate/files/2024-10/SRP-9001-101_English_PLTS.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total, 4 participants were screened for the study. There were no screen failures.
Groups:
- Delandistrogene Moxeparvovec: Participants received a single IV infusion of delandistrogene moxeparvovec on Day 1.
Period: Overall Study
Arm/Group | Delandistrogene Moxeparvovec
Started | 4
Received at Least 1 Dose of Study Drug | 4 (Full Analysis Set)
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: all participants who received study treatment.
Arm/Group | Delandistrogene Moxeparvovec
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.14 (0.91) [lower limit 0.91]
Age, Customized [Number; unit: Participants]
  In utero | 0
  Preterm newborn infants (gestational age < 37 wks) | 0
  Newborns (0-27 days) | 0
  Infants and toddlers (28 days-23 months) | 0
  Children (2-11 years) | 4
  Adolescents (12-17 years) | 0
  Adults (18-64 years) | 0
  From 65-84 years | 0
  85 years and over | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant that does not necessarily have a causal relationship with the study drug. An AE can, therefore, be any unfavorable and unintended symptom, sign, disease, condition, or test abnormality that occurs during or after administration of a study drug, whether or not considered related to the study drug. A summary of serious and all other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Up to 5 years
Population: Full Analysis Set: all participants who received study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Delandistrogene Moxeparvovec
Number analyzed (Participants) | 4
Participants | 4

2. Secondary Outcome: Change From Baseline at Day 90 in Delandistrogene Moxeparvovec Dystrophin Expression as Measured by Western Blot
Description: Baseline muscle biopsies with ultrasound guidance were performed pre-treatment and post-treatment (Day 90) on all participants. The change from baseline in delandistrogene moxeparvovec dystrophin protein levels in these muscle biopsy samples was determined by Western blot. An increase in protein expression indicates production of the delandistrogene moxeparvovec dystrophin protein.
Time Frame: Baseline, Day 90
Population: Full Analysis Set: all participants who received study treatment.
Measure: Mean (Standard Deviation); unit: percent control
Arm/Group | Delandistrogene Moxeparvovec
Number analyzed (Participants) | 4
percent control | 70.52 (76.10) [lower limit 76.10]

3. Secondary Outcome: Change From Baseline at Day 90 in Delandistrogene Moxeparvovec Dystrophin Expression as Measured by Immunofluorescence (IF) Fiber Intensity
Description: Baseline muscle biopsies with ultrasound guidance were performed pre-treatment and post-treatment (Day 90) on all participants. The change from baseline in delandistrogene moxeparvovec dystrophin expression in these muscle biopsy samples was determined using IF. Automated software was used to quantify the intensity of dystrophin expression post-treatment compared to pre-treatment (Percent Normal). The number of muscle fibers expressing micro-dystrophin was quantified by independent trained evaluators. An increase in IF fiber intensity indicates increased delandistrogene moxeparvovec dystrophin expression.
Time Frame: Baseline, Day 90
Population: Full Analysis Set: all participants who received study treatment.
Measure: Mean (Standard Deviation); unit: percent fluorescent expression
Arm/Group | Delandistrogene Moxeparvovec
Number analyzed (Participants) | 4
percent fluorescent expression | 93.59 (43.86) [lower limit 43.86]

4. Secondary Outcome: Change From Baseline at Day 90 in Delandistrogene Moxeparvovec Dystrophin Expression as Measured by IF Percent Dystrophin Positive Fibers (PDPF)
Description: Baseline muscle biopsies with ultrasound guidance were performed pre-treatment and post-treatment (Day 90) on all participants. The change from baseline in delandistrogene moxeparvovec dystrophin expression in these muscle biopsy samples was determined by IF PDPF. Automated software was used to quantify the intensity of dystrophin expression post-treatment compared to pre-treatment (Percent Normal). The number of muscle fibers expressing micro-dystrophin was quantified by independent trained evaluators. An increase in IF PDPF indicates increased delandistrogene moxeparvovec dystrophin expression.
Time Frame: Baseline, Day 90
Population: Full Analysis Set: all participants who received study treatment.
Measure: Mean (Standard Deviation); unit: percent dystrophin positive fibers
Arm/Group | Delandistrogene Moxeparvovec
Number analyzed (Participants) | 4
percent dystrophin positive fibers | 81.18 (10.19) [lower limit 10.19]

5. Secondary Outcome: Change From Baseline at Year 5 in the 100 Meter Timed Test
Description: This assessment measures the time needed to move 100 meters and served as the primary motor outcome measure for this study. A decrease in the time needed to move 100 meters indicates increased motor function.
Time Frame: Baseline, Year 5
Population: Full Analysis Set: all participants who received study treatment.
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Delandistrogene Moxeparvovec
Number analyzed (Participants) | 4
second | -4.02 (4.64) [lower limit 4.64]

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: All reported adverse events are based upon the Full Analysis Set: all participants who received study treatment.
Arm/Group | Delandistrogene Moxeparvovec
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delandistrogene Moxeparvovec (N=4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Asthenia (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (11)
COVID-19 (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (4)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Hepatic enzyme increased (Investigations) | 3 (4)
Influenza A virus test positive (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (3)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Eye irritation (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (15)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Irritability (Psychiatric disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/64/NCT03375164/Prot_000.pdf